CLINICAL TRIAL: NCT01332461
Title: Chronic Obstructive Pulmonary Disease (COPD)-Related Healthcare Utilization and Costs After Discharge From a Hospitalization or Emergency Department Visit on a Regimen of Fluticasone Propionate-Salmeterol Combination Versus Other Maintenance Therapies
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112609
Record Dates: First submitted 2011-03-18; First posted 2011-04-11 (Estimated); Results first posted 2011-04-11 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination; Tiotropium Bromide; Ipratropium; Albuterol, Ipratropium Drug Combination; Salmeterol Xinafoate; Formoterol Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD Patients: Patients over the age of 40 with a COPD-related hospital or ER visit
  Interventions: Drug: fluticasone propionate/salmeterol xinafoate combination; Drug: Other maintenance Treatments (OMT)

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol xinafoate combination — Patients filling a prescription for fluticasone/salmeterol combination as index drug
  Other Names: Advair (TM)
Drug: Other maintenance Treatments (OMT) — OMT group includes tiotropium, ipratropium alone or in combination with albuterol, inhaled steroids, long acting beta agonists
  Other Names: Spiriva (TM); Atrovent (TM); Combivent (TM); Serevent (TM); Foradil (TM)

SUMMARY:
This was a retrospective cross-sectional database study using administrative data (study period: 1/1/2003 through 7/31/2008). Managed care enrollees (aged >40 years) having at least one Hospitalization with primary or secondary diagnosis of COPD (ICD code 491.xx, 492.xx and 496.xx) or at least one Emergency Room (ER) visit with primary diagnosis of COPD (index event) during the study period was the target population. All subjects were required to have one year of pre-index period baseline data. COPD events of interest were ER, Hospital and physician visits followed by oral corticosteroids (OCS) or antibiotics (Ab) within 7 days. Other censoring events were treatment switch; loss of enrollment; >60-day gap between medication fills; or end of study period.

This study is a non descriptive hypothesis testing study. Key study hypotheses are listed below.

Specifically the study hypotheses for the primary outcome being tested were:

Ho: There is no difference in risk of COPD-related hospitalization between FSC and OMT Ha: There is a difference in risk of COPD-related hospitalization between FSC and OMT

Hypothesis for the key secondary outcome of COPD-related costs that was tested was:

Ho: There is no difference in COPD-related costs between FSC and OMT Ha: There is a difference in COPD-related costs between FSC and OMT

ELIGIBILITY:
Inclusion Criteria:

* At least one hospitalization with a primary or secondary diagnosis of COPD or at least one ER visit with a primary diagnosis of COPD
* Initiatiation (prescription) of FSC or non-FSC (i.e. TIO, ICS, LABA, IPR) during peri-index period
* At least 40 years of age
* Continuous eligibility in the pre-index, peri-index, and follow-up periods

Exclusion Criteria

* Presence of exclusionary comorbid conditions during pre-index, peri-index, and follow-up periods: respiratory cancer, cystic fibrosis, fibrosis due to TB, and bronchiectasis, pneumonociosis, pulmonary fibrosis, pulmonary tuberculosis, sarcoidosis
* Controller medication use during peri-index period
* COPD-related hospitalization, ER visit, or physician visit plus OCS/Abx within 3 days of visit during the peri-index period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Managed care enrollees (aged >40 years) having at least one IP with primary or secondary diagnosis of COPD (ICD code 491.xx, 492.xx and 496.xx) or at least one ER visit with primary diagnosis of COPD (index event) during the study period was the target population
Sampling Method: Non-Probability Sample
Enrollment: 5677 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Dalal AA, Shah M, D'Souza AO, Mapel DW. COPD-related healthcare utilization and costs after discharge from a hospitalization or emergency department visit on a regimen of fluticasone propionate-salmeterol combination versus other maintenance therapies. Am J Manag Care. 2011 Mar 1;17(3):e55-65. PMID 21504260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a patient cohort. All diagnoses and treatments are recorded in the course of routine medical practice.
Groups:
- Fluticasone/Salmeterol Combination (FSC) Cohort: Fluticasone/Salmeterol Combination (FSC) 250/50 micrograms (mcg) twice a day
- Other Maintenance Therapies Cohort: Tiotropium, Ipratropium, Ipratropium-albuterol combination drug product, Inhaled corticosteroid, Long-acting beta-agonist. Due to the retrospective nature of this study, dosing information is not available.
Period: Overall Study
Arm/Group | Fluticasone/Salmeterol Combination (FSC) Cohort | Other Maintenance Therapies Cohort
Started | 1291 | 4386
Completed | 1291 | 4386
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone/Salmeterol Combination (FSC) Cohort | Other Maintenance Therapies Cohort | Total
Number analyzed (Participants) | 1291 | 4386 | 5677
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (12.1) | 68.5 (12.1) | 68.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 698 | 2183 | 2881
  Male | 593 | 2203 | 2796

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Having a Hospitalization or Emergency Room (ER) Visit Related to Chronic Obstructive Pulmonary Disease (COPD) Represented Per 100 Person-years
Description: The number of participants (par.) with a COPD-related hospitalization/ ER visit was computed during follow-up (FU) and was standardized by dividing by the total days of FU in each cohort since par. had different lengths of FU. The number of par. per 100 person-years was computed as: numerator = total number of par. with a COPD-related hospitalization/ER visit; denominator = sum of the time of FU in years across all par./100. The index date is defined as the date of discharge from a hospitalization/ER visit for COPD that had a maintenance medication dispensed within 60 days post-discharge.
Time Frame: Maximum of 1 year after index date (Jan 1, 2004 through May 30, 2008)
Population: Managed care enrollees with at least 1 inpatient hospitalization (IP) with primary or secondary diagnosis of COPD (International Classification of Disease (ICD) code 491.xx, 492.xx, and 496.xx) or at least one ER visit with primary diagnosis of COPD during the study period with maintenance medication within 60 days post-discharge
Measure: Number; unit: participants per 100 person-years
Arm/Group | Fluticasone/Salmeterol Combination (FSC) Cohort | Other Maintenance Therapies Cohort
Number analyzed (Participants) | 1291 | 4386
participants per 100 person-years | 8.6 | 16.3
Statistical Analysis 1: Comparison: Fluticasone/Salmeterol Combination (FSC) Cohort vs Other Maintenance Therapies Cohort; Test type: Superiority or Other; p = 0.05, Log Rank; Hazard Ratio (HR) = 0.649, 95% CI 2-sided [0.455 to 0.926] — Covariates for risk models included Charlson Comorbidity Index, presence of asthma, number and quantity of rescue and controller medications, oxygen, and number of COPD healthcare resource use

2. Secondary Outcome: Number of Participants Having a COPD-related Event Related to Chronic Obstructive Pulmonary Disease (COPD) Represented Per 100 Person-years
Description: The number of participants having a COPD-related event was computed during the follow-up and was standardized by dividing by the total days of follow-up in each cohort since patients had different lengths of follow-up. Four types of COPD events were defined: COPD-related hospitalization, emergency room (ER) visit, physician visit with a prescription (Rx) for oral corticosteroid or antibiotic within 3 days of the visit, or combined occurrence of any of the aforementioned three types.
Time Frame: Maximum of 1 year after index date (Jan 1, 2004 through May 30, 2008)
Population: as for outcome 1
Measure: Number; unit: participants per 100 person-years
Arm/Group | Fluticasone/Salmeterol Combination (FSC) Cohort | Other Maintenance Therapies Cohort
Number analyzed (Participants) | 1291 | 4386
participants per 100 person-years
  COPD-related hospitalization | 2.8 | 6.0
  COPD-related ER visit | 6.6 | 12.0
  COPD-related physician + Rx visit | 27.2 | 37.4
  COPD-related hospitalization/ER visit/physician+Rx | 34.6 | 50.7
Statistical Analysis 1: Comparison: Fluticasone/Salmeterol Combination (FSC) Cohort vs Other Maintenance Therapies Cohort; Test type: Superiority or Other; p < 0.05, Log Rank — COPD-related hospitalization; Hazard Ratio (HR) = 0.601, 95% CI 2-sided [0.326 to 1.109] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fluticasone/Salmeterol Combination (FSC) Cohort vs Other Maintenance Therapies Cohort; Test type: Superiority or Other; p < 0.05, Log Rank — COPD-related ER visit; Hazard Ratio (HR) = 0.651, 95% CI 2-sided [0.434 to 0.977] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Fluticasone/Salmeterol Combination (FSC) Cohort vs Other Maintenance Therapies Cohort; Test type: Superiority or Other; p < 0.05, Log Rank — COPD-related physician + Rx visit; Hazard Ratio (HR) = 0.815, 95% CI 2-sided [0.658 to 1.008] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Fluticasone/Salmeterol Combination (FSC) Cohort vs Other Maintenance Therapies Cohort; Test type: Superiority or Other; p < 0.05, Log Rank — COPD-related hospitalization/ER visit/physician+Rx; Hazard Ratio (HR) = 0.785, 95% CI 2-sided [0.649 to 0.948] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Monthly COPD-related Costs Per Participant
Description: Cost categories included medical, pharmacy, and total calculated as the sum of medical and pharmacy. Costs were computed during a variable follow-up period and were standardized on a per-month basis. COPD-related medical costs were computed using claims with a primary diagnosis of COPD, and COPD-related pharmacy costs were computed using the paid amounts of pharmacy claims for prescription medication used for COPD.
Time Frame: Maximum of 1 year after index date (Jan 1, 2004 through May 30, 2008)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States (US) dollars
Arm/Group | Fluticasone/Salmeterol Combination (FSC) Cohort | Other Maintenance Therapies Cohort
Number analyzed (Participants) | 1291 | 4386
United States (US) dollars
  COPD-related total costs | 205 (459.4) | 297 (1376.4)
  COPD-related pharmacy costs | 121 (121.8) | 126 (307.7)
  COPD-related medical costs | 84 (432.5) | 171 (1331.4)

ADVERSE EVENTS:
Description: This study was a retrospective observational study; thus, no serious adverse events or adverse events were collected.
Arm/Group | Fluticasone/Salmeterol Combination (FSC) Cohort | Other Maintenance Therapies Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.